CLINICAL TRIAL: NCT00203801
Title: Open Label Study to Evaluate Combination Anti-malarial Therapy,in Terms of Efficacy, Prevalence of Gametocyte Carriage and Molecular Markers Associated With Sulfadoxine Pyrimethamine Resistance in Uncomplicated Plasmodium Falciparum
Brief Title: Combination Antimalarials in Uncomplicated Malaria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: World Health Organization (Other); Medical Research Council, South Africa (Other); Global Fund (Other)
Responsible Party: Principal Investigator, Professor Karen I Barnes, Professor Karen I Barnes, University of Cape Town
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEACAT 01 Mono (Am 1,2,3,5,6)
Record Dates: First submitted 2005-08-29; First posted 2005-09-20 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Malaria
Keywords: Malaria; Efficacy; Pharmacokinetic; Gametocyte; Molecular markers; Sulfadoxine-pyrimethamine; Artesunate; Artemisinin
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; Artesunate; Artemether, Lumefantrine Drug Combination

INTERVENTIONS:
Drug: Sulfadoxine-pyrimethamine
Drug: Artesunate plus sulfadoxine-pyrimethamine
Drug: Artemether-lumefantrine

SUMMARY:
The purpose of this study is to study the efficacy of sulfadoxine-pyrimethamine on its own and compare this with efficacy of a new combination antimalarial therapy, either sulphadoxine-pyrimethamine plus artesunate or artemether-lumefantrine.

DETAILED DESCRIPTION:
The resistance of Plasmodium falciparum to anti-malarial drugs is a serious impediment to the control of malaria. In the South East African Combination Anti-malarial Therapy (SEACAT) evaluation, there will be a comprehensive evaluation of phased introduction of combination anti-malarials (CAT) in Mozambique, Swaziland and South Africa. In order to facilitate formulation of an effective regional drug policy and provide a database for decision-making on the implementation of combination therapy, it is essential that the in vivo response to CAT in all three countries be investigated. An SP therapeutic efficacy study will be conducted according to this modified World Health Organization (WHO) protocol to guide the selection of CAT. After CAT is introduced an in vivo CAT efficacy study will then be conducted to evaluate the efficacy of artesunate plus SP (or artemether-lumefantrine in KwaZulu Natal and Limpopo). In areas of low intensity malaria transmission the CAT in vivo study results will be compared across sites and with those found at baseline with monotherapy, for each site.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, older than 12 months.
* Weight > 10 kg.
* Diagnoses of uncomplicated acute P. falciparum malaria parasitaemia of up to 250 000 asexual parasite/mcl blood with axillary temperature of greater than and equal to 37.5 or history of fever
* Documented informed consent
* Lives close enough to the health centre for reliable follow up

Exclusion Criteria:

* Has received anti-malarial treatment in the past 7 days.
* Severely ill (based on WHO Criteria for severe malaria ) or if patient is considered, in the opinion of the investigator or designee, to have moderately severe malaria (e.g. prostrate, repeated vomiting, dehydrated).
* Has received cotrimoxazole or chloramphenicol in the past 7 days.
* History of Glucose-6-phosphate dehydrogenase (G6PD) deficiency (not a contra-indication for artemether-lumefantrine).
* Is pregnant or breastfeeding.
* Has a history of allergy to any of the study drugs (including other sulphonamides e.g. cotrimoxazole, other artemisinin derivatives e.g. artemether-lumefantrine).

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 700
Dates: Start 2002-01; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Therapeutic efficacy defined as:
Adequate Clinical and Parasitological Response (ACPR), Early Treatment Failure (ETF), Late Treatment Failure (LTF), defined as Late Clinical Failure (LCF) and Late Parasitological Failure (LPF);
Sensitive or parasitological failure (RI, early and late, RII, RIII)
Parasitological failures will be classified as recrudescence or re-infection (or indeterminate) using glutamate-rich protein (GLURP) and merozoite surface protein (MSP) I & II markers;
Parasite clearance time;
Fever clearance time.

SECONDARY OUTCOMES:
Association between study treatment and gametocyte carriage
Pharmacokinetics by measurement of whole blood levels of Sulfadoxine and Pyrimethamine, and lumefantrine should a reliable assay become available
Correlation of frequency of dihydropteroate synthase (DHFR) and dihydrofolate reductase (DHPS) mutations with parasitological outcome
Tolerability by describing adverse events and changes in haematological parameters
Capacity by describing the training and development of study teams and their subsequent skills attained

CONTACTS AND LOCATIONS:
Overall Officials: Karen Barnes, MBChB, Principal Investigator — University of Cape Town
Locations (7):
- Eswatini (2):
  - Ndzevane Clinic, Ndzevane
  - Vuvulane Clinic, Vuvulane
- Mozambique (2):
  - Bela Vista Clinic, Bela Vista, Matutuine
  - Namaacha Clinic, Namaacha
- South Africa (3):
  - Ndumo Clinic, Ndumo, KwaZulu-Natal
  - Lulekani Clinic, Lulekani, Limpopo
  - Naas Clinic, Naas, Mpumalanga